CLINICAL TRIAL: NCT00859222
Title: Phase I/II Study of LBH589 and Bevacizumab in Patients With Recurrent High Grade Glioma
Brief Title: LBH589 and Bevacizumab in Patients With Recurrent High Grade Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Patrick Y. Wen, MD (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Northwestern University (Other); University of Virginia (Other); Genentech, Inc. (Industry); Novartis (Industry)
Responsible Party: Sponsor-Investigator, Patrick Y. Wen, MD, Director, Center For Neuro-Oncology, Dana-Farber/Brigham and Women's Cancer Center
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-342; CLBH589BUS42T
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Results first posted 2016-11-28 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Malignant Glioma
Keywords: LBH589; bevacizumab; Avastin; Panobinostat
MeSH Terms: conditions — Glioma | interventions — Panobinostat; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Phase I Cohort 1: Bevacizumab +LBH589 20 mg every week (Experimental): Phase I Cohort 1 participants received bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle and the original starting LBH589 dose of 20 mg/day orally, 3x per week, every week (days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26). Participants were treated until disease progression or unacceptable toxicity.
  Interventions: Drug: LBH589; Drug: bevacizumab
- Phase I Cohort 2: Bevacizumab + LBH589 20 mg every other week (Experimental): Phase I Cohort 2 participants received bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle and the amended starting LBH589 dose of 20 mg/day orally, 3x per week, every other week (Days 1, 3, 5, 15, 17, 19). Participants were treated until disease progression or unacceptable toxicity.
  Interventions: Drug: LBH589; Drug: bevacizumab
- Phase I Cohort 3: Bevacizumab + LBH589 30 mg every other week (Experimental): Phase I Cohort 3 participants received bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle and LBH589 30 mg/day orally, 3x per week, every other week (Days 1, 3, 5, 15, 17, 19). Participants were treated until disease progression or unacceptable toxicity.
  Interventions: Drug: LBH589; Drug: bevacizumab
- All Phase I Participants (Experimental): All phase I participants received bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle and LBH589 according to the established dose escalation schedule. Participants were treated until disease progression or unacceptable toxicity.
  Interventions: Drug: LBH589; Drug: bevacizumab
- Phase II GBM: Bevacizumab + LBH589 30 mg every other week (Experimental): Phase II glioblastoma (GBM) participants received the regimen established in the Phase I study (Feb 2011). Phase II participants received bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle and LBH589 30 mg/day orally, 3x per week, every other week (Days 1, 3, 5, 15, 17, 19). Participants were treated until disease progression or unacceptable toxicity.
  Interventions: Drug: LBH589; Drug: bevacizumab
- Phase II AG: Bevacizumab + LBH589 30 mg every other week (Experimental): Phase II Anaplastic Glioma (AG) participants received the regimen established in the Phase I study (Feb 2011). Phase II participants received bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle and LBH589 30 mg/day orally, 3x per week, every other week (Days 1, 3, 5, 15, 17, 19). Participants were treated until disease progression or unacceptable toxicity.
  Interventions: Drug: LBH589; Drug: bevacizumab
- All Phase II Participants (Experimental): All phase II participants received bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle and LBH589 30 mg/day orally, 3x per week, every other week (Days 1, 3, 5, 15, 17, 19). Participants were treated until disease progression or unacceptable toxicity.
  Interventions: Drug: LBH589; Drug: bevacizumab

INTERVENTIONS:
Drug: LBH589
  Other Names: panobinostat; Farydak
Drug: bevacizumab
  Other Names: Avastin

SUMMARY:
The purpose of this research study is to determine the amount of LBH589 that can be given to people safely when LBH589 is given in combination with bevacizumab. LBH589 in combination with bevacizumab is a drug combination that may stop cancer cells from growing abnormally. LBH589 has been used alone in other trials for solid tumor malignancies. Bevacizumab is FDA approved for use in patients with colorectal cancer and has been studied extensively in other types of solid tumors. The combination of LBH589 and bevacizumab has not yet been studied but information from other studies suggests that the combination may help prevent the growth of the participant's tumor.

DETAILED DESCRIPTION:
Phase I

Primary Objective

• To determine the maximum tolerated dose (MTD) of LBH589 in combination with bevacizumab given at 10 mg/kg every 2 weeks in patients with recurrent glioblastoma (GBM), gliosarcoma, anaplastic astrocytoma, anaplastic oligodendroglioma or mixed anaplastic oligoastrocytoma.

Secondary Objective

• To define safety.

Phase II

Primary Objective

• To determine the efficacy of LBH589 in combination with bevacizumab in patients with recurrent GBM or gliosarcoma as measured by 6-month progression-free survival (PFS6).

Secondary Objectives

* To measure overall survival, time-to-tumor progression and objective tumor response.
* To further evaluate safety.

Exploratory Objectives

* To provide preliminary data on the efficacy in patients with recurrent anaplastic astrocytoma, anaplastic oligodendroglioma or mixed anaplastic oligoastrocytoma.
* To explore the relationship of the molecular phenotype of the tumor with survival.
* To investigate correlation of treatment response with laboratory correlates including, plasma angiogenic proteins and perfusion MRI.

Statistical Design

The Phase I study follows a standard 3+3 dose escalation design. Three potential dose levels of oral LBH589 3x per week days 1, 3 and 5 are under evaluation including a starting dose 0 on a weekly schedule as well as dose level 2 and a de-escalation dose level 1 on a weekly schedule. [Note: The study was amended to revise the starting dose due to concerns for thrombocytopenia with the weekly dosing regimen.] The DLT observation period is the first 30 days of treatment. For the Phase II study, based on prior research of bevacizumab monotherapy, a PFS6 rate of 35% does not justify further utilization of LBH589 in combination with bevacizumab while a PFS6 rate of 55% is worthy of further study. With 41 GBM eligible participants in the Phase II study, the treatment would be deemed promising if at least 20 GBM participants achieve 6-month progression-free survival. This design has at least 85% power and a 0.07 significance level to predict the difference between the null hypothesis of 35% PFS6 rate and the alternative hypothesis of 55% PFS6 rate. The protocol specifies a planned interim analysis after the first 21 participants have been accrued. If 12 or more of those participants have died or experienced disease progression/ relapse within 6 months of initiating treatment, accrual will be suspended and the data carefully reviewed before proceeding with additional patient accrual. Participants who are removed from active treatment for toxicity prior to reaching 6 months on treatment are not included in this interim analysis. Participants with recurrent GBM enrolled in the phase I study at the maximum tolerated dose (ie, the phase II dose) are eligible for inclusion in the interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to participation in the study and any related procedures being performed.
* Agreed to and signed an authorization for the release of their protected health information.
* Must be 18 years of age or older
* Karnofsky Performance Status 60 or greater
* Life expectancy of at least 8 weeks
* Histologic diagnosis of GBM, gliosarcoma, anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), or anaplastic mixed oligoastrocytoma (AMO) (Patients are eligible if the original histology was lower-grade glioma)
* Unequivocal progression by magnetic resonance imaging (MRI) or computed tomography (CT) scan. A scan must be performed within 14 days prior to registration and on a steroid dose that has been stable for at least 5 days. (Patients with recurrence who undergo resection and are left without measurable or evaluable disease are eligible.)
* Patients must have failed prior radiation therapy and must have an interval of greater than or equal to 60 days from the completion of radiation therapy to study entry.
* Patients must have recovered from the toxic effects of prior therapy. Residual toxicity from any previous treatment must be Grade 1 or less.
* Sufficient time for recovery from prior therapy: 28 days from any investigational agent, 28 days from prior cytotoxic therapy(except 23 days from prior temozolomide, 14 days from vincristine, 42 days from nitrosoureas, 21 days from procarbazine administration), and 7 days for non-cytotoxic agents.
* Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based upon positron emission tomography (PET), Thallium scanning, MR spectroscopy or surgical documentation of disease.
* Subjects who have undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply: a) prior to initiating therapy, 4 weeks must have elapsed since surgery (Subjects must have recovered from surgical-related trauma. Wound healing needs to have occurred.) b) residual disease following resection of recurrent malignant glioma is not mandated for eligibility. To assess the extent of residual disease postoperatively, a MRI or CT should be done at least 4 weeks postoperatively and within 14 days prior to registration.
* Clinical laboratory tests within 14 days prior to enrollment meeting the criteria listed in the protocol
* Cardiology assessment: Baseline MUGA or Echocardiogram must demonstrate LVEF 50% or greater
* Electrocardiogram: A single screening ECG, taken within 14 days of registration, will be performed to assess study eligibility. Patients whose single QTc interval is ≤ 450 msec are eligible. Patients whose QTc interval is > 460 msec are ineligible. If the result is > 450 msec and ≤ 460 msec, two additional ECG readings are to be performed, each one separated by at least 5 minutes; in this case to be eligible, each individual QTc interval must be ≤ 460 msec and the average of the QTc intervals must be ≤ 450 msec.
* Patient is non-hypertensive or has well-controlled hypertension (systolic blood pressure of < 140mm Hg or diastolic pressure < 90 mm Hg).
* Female subjects of childbearing potential must have a negative pregnancy test confirmed both at screening and within 48 hours prior to dosing with the study drug
* Female subjects of childbearing potential and male subjects with female partner of childbearing potential must agree to use a medically accepted method of contraception while receiving protocol-specified medication, and for 3 months after stopping the medication.
* Subjects must be free of any clinically relevant disease (other than glioma) that would, in the Investigator's opinion, interfere with the conduct of the study or study evaluations.
* Subjects must be able to adhere to the dosing and visit schedules, and agree to record medication times accurately and consistently in a daily diary.

PHASE I Inclusion Criteria (the following modifications to the general eligibility criteria apply to Phase I patients only):

• Patients may have been treated for any number of prior relapses. Relapse is defined as progression following initial therapy

PHASE II Inclusion Criteria (phase II patients must meet the general eligibility criteria as well as the following):

* Patients may have had treatment for no more than 2 prior relapses. (The intent therefore is that patients had no more than 3 prior therapies: initial and treatment for 2 relapses.)
* It is mandatory that 15 unstained paraffin slides or 1 representative tissue block be available from original surgery or definitive surgery or the surgery closest to initiation of this clinical trial.

Exclusion Criteria:

* Subject has received previous therapy with anti-VEGF targeted agents or with any histone deacetylase inhibitors. (Prior treatment with valproic acid for seizures is allowed but requires a washout of at least 14 days prior to starting LBH589.) Although concomitant use of the following drugs is not allowed on study, previous use is allowed, provided patients meet the following mandatory washout periods:

  i. Drugs w/ risk of causing TdP = 72 hrs; ii. Warfarin = 7 days.
* History of grade 2 thrombocytopenia or grade 3 neutropenia on any prior regimen.
* Presence of ≥ grade 2 peripheral neuropathy.
* Bleeding diathesis or coagulopathy
* History of intratumoral or peritumoral hemorrhage if deemed significant by the treating physician
* Treatment with warfarin. (For patients requiring anticoagulation therapy, only therapeutic low molecular weight heparin or factor Xa inhibitors are permitted.)
* Patients who have received any investigational drug or undergone major surgery < 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* Patients with any disease that will obscure toxicity or dangerously alter drug metabolism
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and has not received treatment for that particular disease for a minimum of 3 years
* Impaired cardiac function as detailed in the protocol
* Uncontrolled hypertension (systolic blood pressure >/= 140 mmHg and/or diastolic blood pressure >/= 90 mmHg) and/or prior history of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to Day 1
* Patients with unresolved diarrhea > CTCAE grade 1
* Patients with INR > 1.5
* Patients with major surgery or a significant traumatic injury within 28 days prior to Day 1
* Patients with any condition that impairs their ability to swallow and/or absorb pills
* Concomitant use of drugs with a risk of causing torsades de pointes
* Concomitant use of CYP3A4 inhibitors during the treatment phase of the study and within 72 hours prior to starting treatment
* Concomitant use of potent CYP3A4/5 inducers during the treatment phase of the study and within 2 weeks prior to starting treatment
* Concomitant use of any anti-cancer therapy or radiation therapy, or any other investigational agent
* Patients has known human immunodeficiency virus (HIV) of hepatitis C infection (baseline testing for HIV or hepatitis C is not required)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to LBH589 or bevacizumab, or their excipients
* Patient is in a situation or condition that, in the opinion of the investigator, may interfere with optimal participation in the study
* Patient has a significant history of non-compliance to medical regimens
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria as demonstrated by a UPC ratio of 1.0 or greater at screening
* Subject is pregnant or intends to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-03; Primary Completion 2013-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y. Wen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth-Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Virginia, Department of Neurology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Drappatz J, Lee EQ, Hammond S, Grimm SA, Norden AD, Beroukhim R, Gerard M, Schiff D, Chi AS, Batchelor TT, Doherty LM, Ciampa AS, Lafrankie DC, Ruland S, Snodgrass SM, Raizer JJ, Wen PY. Phase I study of panobinostat in combination with bevacizumab for recurrent high-grade glioma. J Neurooncol. 2012 Mar;107(1):133-8. doi: 10.1007/s11060-011-0717-z. Epub 2011 Oct 8. PMID 21984064
- [Result] Lee EQ, Reardon DA, Schiff D, Drappatz J, Muzikansky A, Grimm SA, Norden AD, Nayak L, Beroukhim R, Rinne ML, Chi AS, Batchelor TT, Hempfling K, McCluskey C, Smith KH, Gaffey SC, Wrigley B, Ligon KL, Raizer JJ, Wen PY. Phase II study of panobinostat in combination with bevacizumab for recurrent glioblastoma and anaplastic glioma. Neuro Oncol. 2015 Jun;17(6):862-7. doi: 10.1093/neuonc/nou350. Epub 2015 Jan 7. PMID 25572329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in the Phase I study enrolled from March 2009-January 2011 and the Phase II study from June 2011-May 2013.
Period: Overall Study
Arm/Group | Phase I Cohort 1: Bevacizumab +LBH589 20 mg Every Week | Phase I Cohort 2: Bevacizumab + LBH589 20 mg Every Other Week | Phase I Cohort 3: Bevacizumab + LBH589 30 mg Every Other Week | Phase II GBM: Bevacizumab + LBH589 30 mg Every Other Week | Phase II AG: Bevacizumab + LBH589 30 mg Every Other Week
Started | 3 | 3 | 6 | 24 | 15
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 6 | 24 | 15
Not completed — Adverse Event | 2 | 3 | 6 | 24 | 15
Not completed — DLT | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled patients.
Groups:
- All Phase I Participants: All phase I participants received bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle and LBH589 according to the established dose escalation schedule.
- Total: Total of all reporting groups
Arm/Group | All Phase I Participants | Phase II GBM: Bevacizumab + LBH589 30 mg Every Other Week | Phase II AG: Bevacizumab + LBH589 30 mg Every Other Week | Total
Number analyzed (Participants) | 12 | 24 | 15 | 51
Age, Continuous [Median (Full Range); unit: years] | 50 [30 to 71] | 53 [22 to 66] | 48 [31 to 69] | 50 [22 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 5 | 21
  Male | 6 | 14 | 10 | 30
Race/Ethnicity, Customized [Number; unit: participants]
  White | 12 | 16 | 14 | 42
  Non-White | 0 | 8 | 1 | 9
Number of Prior Relapses [Number; unit: participants]
  1 | 12 | 15 | 7 | 34
  2 | 0 | 9 | 4 | 13
  3 | 0 | 0 | 3 | 3
  4 | 0 | 0 | 1 | 1
Histology [Number; unit: participants]
  glioblastoma (GBM) | 10 | 24 | 0 | 34
  anaplastic astrocytoma (AA) | 1 | 0 | 8 | 9
  anaplastic oligodendroglioma (AO) | 0 | 0 | 5 | 5
  anaplastic oligoastrocytoma (AOA) | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: LBH589 Maximum Tolerated Dose (MTD) [Phase I]
Description: The MTD LBH589 in combination with bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle is determined by the number of patients who experience a dose limiting toxicity (DLT). See subsequent primary outcome measure for the DLT definition. The MTD is defined as the highest dose at which fewer than one-third of patients experience a DLT. If no DLTs are observed, the MTD is not reached but the highest dose received may be the Recommended Phase II Dose (RP2D). The MTD was not reached with 0 of 6 DLTs observed in the highest dose cohort but due to safety concerns higher doses of LBH589 with bevacizumab were neither planned nor tested. The RP2D was 30 mg/day orally, 3x per week, every other week.
Time Frame: Participants were assessed every 2 weeks while on study; The observation period for MTD evaluation was the first 30 days of treatment.
Population: All PI participants who received at least one dose of the study drug were evaluable for MTD.
Measure: Number; unit: mg/day orally, 3x per wk, every other wk
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 12
mg/day orally, 3x per wk, every other wk | 30

2. Primary Outcome: Dose Limiting Toxicity (DLT) [Phase I]
Description: A DLT was defined as an adverse event that (a) is related to the LBH589 and/or bevacizumab with an attribution of possible, probable, or definite, and (b) occurs during and/or begins during the first 30 days of the study treatment, and (c) meets any of the following criteria: grade 3 thrombocytopenia; grade 4 neutropenia lasting 7 days; grade 4 anemia lasting 7 days despite transfusion or growth factors; febrile neutropenia if ANC<0.5 x10^9/L; a QT interval corrected for heart rate (QTc) of 500-515 msec that did not stabilize to <480 msec after one week; a second occurrence of QTc 500-515 msec; any QTc >515 msec; any deep vein thrombosis (DVT) or pulmonary embolism (PE) while on fully therapeutic anticoagulation therapy; Grade 3 proteinuria lasting 14 days; or any other clinically significant Grade 3 toxicity despite maximal medical therapy lasting 7 days, any Grade 4 toxicity despite maximal medical therapy; or any Grade 3 or 4 toxicity resulting in study drug discontinuation.
Time Frame: Participants were assessed every 2 weeks while on study; The observation period for DLT evaluation was the first 30 days of treatment.
Population: All PI participants who received at least one dose of the study drug were evaluable for DLT.
Measure: Number; unit: participants with DLT
Arm/Group | Phase I Cohort 1: Bevacizumab +LBH589 20 mg Every Week | Phase I Cohort 2: Bevacizumab + LBH589 20 mg Every Other Week | Phase I Cohort 3: Bevacizumab + LBH589 30 mg Every Other Week
Number analyzed (Participants) | 3 | 3 | 6
participants with DLT | 1 | 0 | 0

3. Primary Outcome: 6-Month Progression-Free Survival (PFS6) [Phase II]
Description: PFS6 is the proportion of patients remaining alive and progression-free at 6-months from study entry. Progressive disease was established based on RANO criteria (Wen et al JCO 2010).
Time Frame: Disease was assessed radiographically to document clinical progression every cycle on treatment and post-treatment every 8 weeks up to 12 months. Participants were followed for PFS6 up to 6 months since study entry.
Population: All participants with measurable disease present at baseline and received at least one dose of the study drug were evaluable for PFS6.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase II GBM: Bevacizumab + LBH589 30 mg Every Other Week | Phase II AG: Bevacizumab + LBH589 30 mg Every Other Week
Number analyzed (Participants) | 24 | 15
proportion of participants | 0.304 [0.124 to 0.507] | 0.467 [0.21 to 0.73]

4. Secondary Outcome: Best Radiographic Response
Description: Radiographic response was established based on Response Assessment in Neuro-Oncology (RANO) criteria (Wen et al JCO 2010) with 5 potential categories: Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive disease (PD) and Unknown status.
Time Frame: Disease was assessed radiographically for response every cycle on treatment. Treatment duration in cycles was a median (range) of 2 (1-6) PI Cohort 1, 4.5 (2-6) PI Cohort 2, 6 (2-10) PI Cohort 3, 5 PII GBM and 7 PII AG.
Population: All participants with measurable disease present at baseline and received at least one dose of the study drug were evaluable for response.
Measure: Number; unit: participants
Arm/Group | Phase I Cohort 1: Bevacizumab +LBH589 20 mg Every Week | Phase I Cohort 2: Bevacizumab + LBH589 20 mg Every Other Week | Phase I Cohort 3: Bevacizumab + LBH589 30 mg Every Other Week | Phase II GBM: Bevacizumab + LBH589 30 mg Every Other Week | Phase II AG: Bevacizumab + LBH589 30 mg Every Other Week
Number analyzed (Participants) | 3 | 3 | 6 | 24 | 15
participants
  Complete Response | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 1 | 2 | 7 | 4
  Stable Disease | 2 | 2 | 3 | 14 | 9
  Progressive Disease | 1 | 0 | 1 | 3 | 2

5. Secondary Outcome: Progression-Free Survival (PFS) [Phase II]
Description: PFS is defined as the time from study entry to the earliest documentation of disease progression or death. Patients alive without evidence of PD were censored at the date of last disease assessment.
Time Frame: Disease was assessed radiographically to document clinical progression every cycle on treatment and post-treatment every 8 weeks up to 12 months.
Population: All PII participants with measurable disease present at baseline and received at least one dose of the study drug were evaluable for PFS.
Measure: Median (Full Range); unit: months
Arm/Group | Phase II GBM: Bevacizumab + LBH589 30 mg Every Other Week | Phase II AG: Bevacizumab + LBH589 30 mg Every Other Week
Number analyzed (Participants) | 24 | 15
months | 5 [3 to 9] | 7 [2 to 10]

6. Other Pre Specified Outcome: Progression-Free Survival (PFS) [Phase I]
Description: PFS is defined as the time from study entry to the earliest documentation of disease progression or death. Patients alive without evidence of PD were censored at the date of last disease assessment. Progressive disease was established based on Response Assessment in Neuro-Oncology (RANO) criteria (Wen et al JCO 2010).
Time Frame: as for outcome 5
Population: All participants with measurable disease present at baseline and received at least one dose of the study drug were evaluable for PFS.
Measure: Median (Full Range); unit: months
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 12
months | 4.3 [1.1 to 9.5]

7. Other Pre Specified Outcome: 6-Month Progression-Free Survival (PFS6) [Phase I]
Description: PFS6 is the proportion of patients remaining alive and progression-free at 6-months from study entry. Progressive disease was established based on Response Assessment in Neuro-Oncology (RANO) criteria (Wen et al JCO 2010).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 12
proportion of participants | 0.25 [0.063 to 0.551]

8. Secondary Outcome: Overall Survival [Phase II]
Description: OS is defined as the time from study entry to death or date last known alive.
Time Frame: Participants were followed long-term for survival every 4 months from the end of treatment until death or lost to follow-up. Phase II participants were followed for OS up to 27 months on this study.
Population: All participants who received at least one dose of the study drug were followed for OS.
Measure: Median (Full Range); unit: months
Arm/Group | Phase II GBM: Bevacizumab + LBH589 30 mg Every Other Week | Phase II AG: Bevacizumab + LBH589 30 mg Every Other Week
Number analyzed (Participants) | 24 | 12
months | 9 [6 to 19] | 17 [5 to 27]

9. Other Pre Specified Outcome: Overall Survival (OS) [Phase I]
Description: OS is defined as the time from study entry to death or date last known alive.
Time Frame: Participants were followed long-term for survival every 4 months from the end of treatment until death or lost to follow-up. Phase I participants were followed for OS up to 12.1 months on this study.
Population: All participants who received at least one dose of the study drug were followed for OS.
Measure: Median (Full Range); unit: months
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 12
months | 8.2 [4.8 to 12.1]

ADVERSE EVENTS:
Time Frame: Assessed each treatment cycle from time of first dose and up to day 30 post-treatment. Treatment duration in cycles was a median (range) of 2 (1-6) Phase I Cohort 1, 4.5 (2-6) Phase I Cohort 2, 6 (2-10) Phase I Cohort 3, 5 Phase II GBM and 7 Phase II AG.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with LBH589 and/or bevacizumab treatment-attribution of at least possibly and grade 3 or higher per CTCAEv3. Other AEs were defined as events with LBH589 and/or bevacizumab treatment-attribution of at least possibly and grades 1 or 2 per CTCAEv3.
Arm/Group | Phase I Cohort 1: Bevacizumab +LBH589 20 mg Every Week | Phase I Cohort 2: Bevacizumab + LBH589 20 mg Every Other Week | Phase I Cohort 3: Bevacizumab + LBH589 30 mg Every Other Week | Phase II GBM: Bevacizumab + LBH589 30 mg Every Other Week | Phase II AG: Bevacizumab + LBH589 30 mg Every Other Week
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 2/6 | 12/24 | 7/15
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 21/24 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Cohort 1: Bevacizumab +LBH589 20 mg Every Week (N=3) | Phase I Cohort 2: Bevacizumab + LBH589 20 mg Every Other Week (N=3) | Phase I Cohort 3: Bevacizumab + LBH589 30 mg Every Other Week (N=6) | Phase II GBM: Bevacizumab + LBH589 30 mg Every Other Week (N=24) | Phase II AG: Bevacizumab + LBH589 30 mg Every Other Week (N=15)
ADH secretion abnormality (eg SIADH) (Investigations) | 0 | 0 | 0 | 1 | 0
ALT, SGPT (Investigations) | 0 | 0 | 0 | 2 | 0
CNS, hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Esophagus, hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1
Head/headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hematologic-other (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 2
Lymphopenia (Investigations) | 0 | 0 | 1 | 2 | 1
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Neutrophils (Investigations) | 0 | 0 | 0 | 2 | 1
Platelets (Investigations) | 1 | 0 | 0 | 3 | 3
QTc interval (Investigations) | 0 | 0 | 1 | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1 | 0 | 4 | 0
Weight loss (Investigations) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Cohort 1: Bevacizumab +LBH589 20 mg Every Week (N=3) | Phase I Cohort 2: Bevacizumab + LBH589 20 mg Every Other Week (N=3) | Phase I Cohort 3: Bevacizumab + LBH589 30 mg Every Other Week (N=6) | Phase II GBM: Bevacizumab + LBH589 30 mg Every Other Week (N=24) | Phase II AG: Bevacizumab + LBH589 30 mg Every Other Week (N=15)
Abdomen, pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Alkaline phosphatase (Investigations) | 1 | 0 | 1 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0
ALT, SGPT (Investigations) | 0 | 0 | 3 | 2 | 6
Amylase (Investigations) | 0 | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4 | 3
Anus, hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
AST, SGOT (Investigations) | 1 | 0 | 4 | 4 | 4
Bicarbonate (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 1
Cardiac-ischemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
CNS, hemorrhage (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Constitutional, other (General disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Creatinine (Investigations) | 1 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 0 | 1 | 5 | 14 | 10
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dry eye syndrome (Eye disorders) | 0 | 0 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Edema limb (General disorders) | 0 | 0 | 0 | 1 | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 4 | 14 | 7
Febrile neutropenia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
GI-other (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 2
Head/headache (Nervous system disorders) | 1 | 0 | 0 | 2 | 1
Hemoglobin (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2 | 3
Hemorrhage-other (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hyopthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Hyopthyroidism (Endocrine disorders) | 0 | 0 | 0 | 2 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 1
Hypertension (Vascular disorders) | 1 | 1 | 2 | 4 | 6
Hyperthyroidism, thyrotoxicosis (Endocrine disorders) | 0 | 0 | 2 | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Infection Gr0-2 neut, vagina (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Infection-other (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Irregular menses (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3 | 1
Leak, CSF (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Leukocytes (Investigations) | 2 | 0 | 4 | 3 | 6
Lipase (Investigations) | 0 | 0 | 0 | 0 | 1
Lymphopenia (Investigations) | 0 | 0 | 0 | 1 | 2
Metabolic/Laboratory-other (Investigations) | 0 | 0 | 0 | 0 | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Muscle, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 5 | 5
Neck, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Neutrophils (Investigations) | 2 | 0 | 4 | 2 | 6
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 4 | 3
Oral cavity, hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pain-other (General disorders) | 0 | 0 | 1 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Platelets (Investigations) | 2 | 0 | 5 | 7 | 6
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
QTc interval (Investigations) | 0 | 0 | 1 | 0 | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin-other (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 0
Speech impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Taste disturbance (Nervous system disorders) | 0 | 0 | 1 | 3 | 4
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 6 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 3
Weight loss (Investigations) | 0 | 0 | 0 | 2 | 0
Wound - non-infectious (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No